CLINICAL TRIAL: NCT01756365
Title: Autologous Cultured Corneal Epithelium ( Culture d'épithélium cornéen Autologue CECA) for the Treatment of Unilateral Corneal Lesions Associated With Limbal Stem Cell Deficiency
Brief Title: Autologous Cultured Corneal Epithelium (CECA) for the Treatment of Limbal Stem Cell Deficiency
Acronym: CECA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Responsible Party: Principal Investigator, Ralph Kyrillos, Principal Investigator, CHU de Quebec-Universite Laval
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LOEX 015
Record Dates: First submitted 2012-12-20; First posted 2012-12-25 (Estimated); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Limbal Stem Cell Deficiency
MeSH Terms: conditions — Limbal Stem Cell Deficiency

STUDY DESIGN:
Intervention Model Description: The culture of corneal epithelium strives to produce a reconstructed tissue with the therapeutical aim of treatment of limbal stem cell deficiency. The study is a phase I / phase II study with the goal to evaluate safety and efficacy of the CECA graft for the treatment of human patients suffering from limbal stem cell deficiency.
Oversight: Data Monitoring Committee: No

ARMS (1):
- ACCE (Autologous Cultured Corneal Epithlium) graft for the treatment of corneal lesions (Experimental): Surgical transplantation of Autologous Cultured Corneal Epithelium
  Interventions: Procedure: Surgical transplantation of ACCE

INTERVENTIONS:
Procedure: Surgical transplantation of ACCE — The culture of corneal epithelium strives to produce a reconstructed tissue with the therapeutical aim of treatment of limbal stem cell deficiency.

SUMMARY:
The study " Autologous cultured corneal epithelium (CECA) for the treatment of corneal lesions associated with limbal stem cell deficiency" is the first clinical trial of this product manufactured at the LOEX laboratory. The culture of corneal epithelium strives to produce a reconstructed tissue with the therapeutical aim of treatment of limbal stem cell deficiency. The study is a phase I/phase II study with the goal to evaluate safety and efficacy of the CECA graft for the treatment of human patients suffering from limbal stem cell deficiency.

The trial is open to all genders. The inclusion of 5 minors is planned.

ELIGIBILITY:
Inclusion Criteria:

All genders

* Adults
* Minors
* LSCD in one or two eyes. A minimum of 1-3 mm2 of undamaged limbus is required for a biopsy to be taken without foreseeable adverse consequences for the donor eye

Exclusion Criteria:

* Donor eye not sufficiently healthy to allow for the harvesting of a 1-3 mm2 limbal biopsy without foreseeable consequences for the donor eye
* Pregnancy
* Breast-feeding
* Incapacitated person
* known allergy to aprotinine (Trasylol (R))
* Hypersensibility to bovine proteins

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2012-12; Primary Completion 2025-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Anatomic assessment | 1 year
  Global severity score (Epithelial deficit, corneal opacity, peripheral and central vascularization, integrity of the ocular surface)

SECONDARY OUTCOMES:
Best corrected visual acuity | 1 year
  Evaluation according to Snellen chart
Level of pain | 1 year
  11 point numerical verbal scale
Quality of life measurements | 1 year
  Health Utilities Index Mark 3

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Kyrillos, MD FRCS (C), Principal Investigator — CHU de Quebec
Locations (4):
- Canada (4):
  - University Health Network - Toronto Western Hospital, Toronto, Ontario
  - CIUSSS de l'Est de l'île de Montréal, Montreal, Quebec
  - McGill University Health Centre; Centre de Médecine Innovatrice/Centre for Innovative Medicine, Montreal, Quebec
  - Centre universitaire d'Ophtalmologie CHU de Québec - HSS, Québec, Quebec